CLINICAL TRIAL: NCT02352623
Title: Quality of Life and Surgical Late Effects of Melanoma Treatment
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, caroline gjørup, M.D. ph.d. student, Herlev Hospital
Other Study IDs: H-4-2014-127
Record Dates: First submitted 2015-01-19; First posted 2015-02-02 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Melanoma; Quality of Life; Lymphedema; Depression; Anxiety; Pain; Cicatrix
MeSH Terms: conditions — Melanoma; Lymphedema; Depression; Anxiety Disorders; Pain; Cicatrix | interventions — Absorptiometry, Photon; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cutaneous melanoma AJCC stage IB-III: Patients treated for cutaneous melanoma (AJCC stage IB-III) will fill out a questionnaire, undergo clinical examination and DXA scan
  Interventions: Radiation: DXA scan; Procedure: Clinical examination

INTERVENTIONS:
Radiation: DXA scan — DXA scan
Procedure: Clinical examination — Clinical examination

SUMMARY:
Health-related Quality of life in Danish stage IB-III cutaneous melanoma patients.

DETAILED DESCRIPTION:
The aim of the PhD-study is to evaluate, in a large cohort of Danish melanoma patients:

1. Health-related quality of life assessing psychological, physical and social well-being
2. Physical long term side effects (lymphoedema, scarring and neuropathic pain)
3. Lymphoedema assessed by clinical examination and DXA scans

ELIGIBILITY:
Inclusion Criteria:

* AJCC stage IB-III cutaneous melanoma patients
* At least one year follow-up after melanoma surgery

Exclusion Criteria:

* Pregnancy
* Bilateral axilla or groin melanoma surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for cutaneous melanoma (AJCC stage IB-III) with wide local excision (WLE) and sentinel lymph node biopsy (SNB) and/ or complete lymph node dissection in the axilla and/or groin will be included in the study.
Sampling Method: Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Global Health Score | 12 months
  Quality of life will be assessed with the questionnaire EORTC QLQ-C30 v.3.0

SECONDARY OUTCOMES:
Anxiety | 12 months
  Anxiety will be assessed with the questionnaire Hospital Anxiety and Depression Scale (HADS)
Depression | 12 months
  Depression will be assessed with the questionnaire Hospital Anxiety and Depression Scale (HADS)
Lymphoedema | 12 months
  Lymphoedema will be assessed with a questionnaire including the LYMQOL questionnaire, clinical examination and DXA scan
Neuropathic pain | 12 months
  Neuropathic pain will be assessed with a questionnaire including painDetect
Volume and tissue composition assessed with DXA scan | 12 months
  DXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Asirvatham Gjørup, MD, Principal Investigator — Department of Plastic Surgery
Locations (1):
- Department of Plastic Surgery, Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gjorup CA, Groenvold M, Hendel HW, Dahlstroem K, Drzewiecki KT, Klausen TW, Holmich LR. Health-related quality of life in melanoma patients: Impact of melanoma-related limb lymphoedema. Eur J Cancer. 2017 Nov;85:122-132. doi: 10.1016/j.ejca.2017.07.052. Epub 2017 Sep 15. PMID 28918186